CLINICAL TRIAL: NCT07330765
Title: Analgesic Efficacy of Pre-Operative Dose of Palmitoylethanolamide in Patients Undergoing Total Knee Arthroplasty, A Randomized Double-Blinded Controlled Trial.
Brief Title: Analgesic Efficacy of Pre-Operative Dose of Palmitoylethanolamide in Patients Undergoing Total Knee Arthroplasty
Acronym: Total knee
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abdelrahman Gaber Sayed Elkhateeb (Other)
Responsible Party: Sponsor-Investigator, Abdelrahman Gaber Sayed Elkhateeb, Assistant lecturer, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pain antieffect of PEA in TKR
Record Dates: First submitted 2025-09-27; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Total Knee Replacement
Keywords: Post operative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo effect on post operative pain after TKA (Experimental): The patient will be gaven an empty pill and we will score the pain postoperative and if it has effect on postoperative pain or not
  Interventions: Drug: Effect of two different drugs on post operative pain after TKA
- Palmetoyelethenolamide effect on post operative pain after TKA (Experimental): The patient will be gaven an pill containing palmytoiethenolamide and we will score the pain postoperative and if it has effect on postoperative pain or not
  Interventions: Drug: Effect of two different drugs on post operative pain after TKA

INTERVENTIONS:
Drug: Effect of two different drugs on post operative pain after TKA — Effect of preoperative dose of palmetoyelethenolamide in post-op pain in patient undergoing Total Knee Replacement
  Other Names: Palmetoyelethenolamide; Placebo pill

SUMMARY:
Analgesic Efficacy of Pre-Operative Dose of palmitoylethanolamide in Patients Undergoing total Knee Arthroplasty, A Randomized Double-Blinded Controlled Trial.

DETAILED DESCRIPTION:
Elective total knee arthroplasty (TKA) is the gold standard for management of arthritis-associated pain and disability in osteoarthritis patients who have failed non-operative treatment modalities Following TKA, patients experience severe pain mediated by multiple pathways Painful stimuli to the body are detected by the free endings of peripheral nerves called nociceptors . Pre-emptive analgesia is analgesia given before the onset of painful stimuli to prevent central sensitization of nervous system to subsequent stimuli that could increase pain Studies have shown that pre-emptive analgesia reduce immediate postoperative pain and also prevent the development of chronic pain by decreasing altered sensory processing .

Multi-modal analgesia is the rational approach to pain management since no single analgesia targets all types of pain

. Increasing evidence has shown that neuro-inflammation plays a key role in pain progression which is sustained by an imbalance within pro-inflammatory and pro-resolving mediators Acylethanolamines (NAEs) are a family of endogenous bio active lipids that regulate multiple processes including pain and inflammation . One of the most widely studied NAEs is the analgesic endocannabinoid compound, palmitoylethanolamide (PEA). Previous research has demonstrated the effectiveness of PEA on conditions characterized by chronic and/or neurological pain The aim of the study is to investigate the safety, tolerability and efficacy of doses of PEA on symptoms of post operative pain.

ELIGIBILITY:
Inclusion Criteria:

Patients Undergoing Total Knee Replacement from 40 years old to 80 years old

Exclusion Criteria

* Rheumatoid Arthritis

  * History of Renal impairment
  * Any complications of surgery as( iatrogenic fractures -patient with low bone quality that needs long stem prosthesis -patient with depressed tibial plateau that needs graft )
  * Patients refused to be enrolled in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2027-10-13 (Estimated); Study Completion 2027-10-13 (Estimated)

PRIMARY OUTCOMES:
Decrease post operative pain | Frist 24 hours postoperative
  Visual Analog Scale (VAS) will be used at 6, 12, 24 hours post-surgery for assessment of Pain. Scale from one to ten Ten means patient in sever pain One means patient is well The higher the score the pain is severer

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
It's an experimental study it will be shared if the outcomes of the study are valid to be shared

REFERENCES:
- [Result] https://pmc.ncbi.nlm.nih.gov/articles/PMC10053226/#:~:text=Palmitoylethanolamide%20(PEA)%2C%20a%20naturally,pain%2C%20although%20this%20remains%20controversial
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/24952959/
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC7132032/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22697514/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37883429/